CLINICAL TRIAL: NCT05450068
Title: Effects of Combining Mobilization With Movement and Spencer's Technique in Diabetic Adhesive Capsulitis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/1012 Bushra
Record Dates: First submitted 2022-04-09; First posted 2022-07-08 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Adhesive Capsulitis
MeSH Terms: conditions — Bursitis | interventions — Movement

STUDY DESIGN:
Who Masked: Participant
Masking Description: Study is single-blinded as the participants are unaware of the treatment given to them.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A-Combined Group (Active Comparator): Participants in this group will receive both Mulligan's mobilization with movement and Spencer's muscle energy technique along with conventional therapy and home exercise plan. 3 sessions per week will be given for 4 weeks.
  Interventions: Other: Mulligan's Mobilization with movement; Other: Spencer's muscle energy technique; Other: Conventional Therapy
- Group B-Mulligan Group (Active Comparator): Participants in this group will receive Mulligan's mobilization with movement along with conventional therapy and home exercise plan. 3 sessions per week will be given for 4 weeks.
  Interventions: Other: Mulligan's Mobilization with movement
- Group C-Spencer Group (Active Comparator): Participants in this group will receive Spencer's muscle energy technique along with conventional therapy and home exercise plan. 3 sessions per week will be given for 4 weeks.
  Interventions: Other: Spencer's muscle energy technique
- Group D-Conventional Group (Active Comparator): Participants in this group will receive conventional therapy alone in hospital with home exercise plan. 3 sessions per week will be given for 4 weeks.
  Interventions: Other: Conventional Therapy

INTERVENTIONS:
Other: Mulligan's Mobilization with movement — The Mulligan's technique will be performed as described by Brian Mulligan. 3 sets of 10 repetitions with 1 minute rest between sets.
  Arms: Group A-Combined Group; Group B-Mulligan Group
Other: Spencer's muscle energy technique — Muscle energy technique that is composed of 7 stages repeated on after the other will be performed. Each movement will be repeated 10 times with 1 minute rest between each set.
  Arms: Group A-Combined Group; Group C-Spencer Group
Other: Conventional Therapy — Electrotherapy-Ultrasound (5-10 mins), Exercise therapy program (isometric, capsular stretching, pectoral stretch and scapular stabilization exercises)
  Arms: Group A-Combined Group; Group D-Conventional Group

SUMMARY:
This study will be a randomized control trial conducted on 44 patients diagnosed as adhesive capsulitis in headquarter hospital Gujar khan. Subjects will be divided equally into 4 groups (n=11 in each group) that are Group A, B, C and D by sealed envelope method. Pre-intervention assessment will be done by using data collection tools and then intervention will be applied. Group A will receive mobilization with movement (MWM) technique along with Spencer's muscle energy technique (MET) with conventional therapy. Group B will receive MWM along with conventional therapy. Group C will receive Spencer's MET along with conventional therapy. Group D will receive conventional therapy alone. All subjects will be given a home exercise plan. Assessment will be done after 1st session, 1st week, 2nd week, 3rd week and finally after 2 weeks on follow up using data collection tool. Data collection tools are semi-structured questionnaire (informed consent, demographic details, goniometric measurements), Visual analogue scale (VAS), shoulder pain and disability index (SPADI) and universal goniometer.

DETAILED DESCRIPTION:
One of the numerous disorders that causes pain and increase resistance to the active and passive movements of shoulder is the adhesive capsulitis. The pathology of the shoulder can be the extrinsic or intrinsic that induces pain and stiffness that is why the treatment should be according to the actual cause of pathology. Another term which is used for these pathology is 'Frozen Shoulder' which is used by the Codman for the first time in history. Adhesive capsulitis does not represent a single pathology rather it is applicable to most of the conditions that causes myospasm most specifically adhesion that forms in the bursa or joint capsule and rotators of the shoulder. Most specifically the term adhesive capsulitis is actually a pathology that includes the capsule's inflammation which results in thickness and fibrosis and consequently adherence to the shoulder as well as the neck of humerus.

About 2%-5% of the global population is affected by the adhesive Capsulitis that's why it is considered as a common condition. Frozen shoulder the alternative term for adhesive capsulitis affect the 2% of the total world population because of the absent of most accurate criteria for diagnosis and sometime due to the over diagnosis. It is uncommon in people under the age of 40, peak prevalence is in people elder than 40 and younger than 60 and is uncommon in people above 70years except for secondary cause and in the manual workers as according to a cumulative incidence of 2.4 persons per 1000 in a year. Economically the impact of adhesive Capsulitis is underscored i-e 8.2% for men and 10.1% for women for adults in working age. It is more prevalent in women as compared to the men. It cannot develop in the same shoulder after the first time but in 20% of people it is seen to develop in the opposite Shoulder.14% of patients have seen to develop in both shoulders at one time, and 80% are those who develop this condition on opposite side within the next five years.

Frozen shoulder is mostly common in patients suffering from diabetes mellitus. 71.5% of the people are estimated to have the diabetes and frozen shoulder at the same time half of them are previously diagnosed with type I or type II diabetes mellitus and remaining have high glucose tolerance test or increased fasting glucose level.The suspected risk of having frozen shoulder have increased a 10% to 20% in people who are diabetic, having 4% point prevalence, and 2-4 times on greater risk as compared to normal population.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female
* Age bracket is 30-70 years
* Pain in the shoulder for at least three months
* All active and passive shoulder movements restricted, with a reduction in external rotation of at least 50%.

Exclusion Criteria:

* Patients with

  * Recent history of surgery on particular shoulder
  * Post-traumatic and rotator cuff rupture
  * Neurological deficits affecting shoulder function
  * Pain or disorders of cervical spine, elbow, wrist or hand
  * Tendon calcification
  * Rheumatoid arthritis
  * Osteoporosis
  * Malignancies
  * Pregnancy
  * Open wounds or skin infections
  * Recent steroid injection
  * Previous manipulation under anesthesia of affected shoulder.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | 6th week.
  A Visual Analogue Scale (VAS) is one of the pain rating scales used for measurement of pain intensity. The findings suggested that 100-mm VAS ratings of 0 to 4 mm can be considered no pain; 5 to 44 mm, mild pain; 45 to 74 mm, moderate pain; and 75 to 100 mm, severe pain. It will be used at baseline, after first session and then every week up to 6th week.
Shoulder Pain and Disability Index | 6th week
  The Shoulder Pain and Disability Index (SPADI) is a patient completed questionnaire with 13 items assessing pain level and extent of difficulty with Activity of daily Livings requiring the use of the upper extremities. The pain subscale has 5-items and the Disability subscale has 8-items.
  It will be used at baseline, every week up to 4th week and then after 2 week follow up on 6th week
Range of Motion | 6th week.
  Ranges of motions of all shoulder movements will be measured. These include Flexion, Abduction, Eternal and Internal Rotation. It will be measured at baseline, after first session, every week up to 4th week and then after 2 week follow up on 6th week.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Khalid, MSOMPT, Principal Investigator — Riphah International University
Locations (1):
- Tehsil headquarter hospital, Gujar Khān, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No